CLINICAL TRIAL: NCT06486090
Title: Effectiveness and Process Evaluation of the Injury-preventive Program #Utviklingsklar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Linkoeping University (Other Government); University of Bath (Other); The Norwegian Olympic and Paralympic Committee and Confederation of Sports (Unknown); The Norwegian Football Federation (Unknown); The Norwegian Handball Federation (Unknown)
Responsible Party: Principal Investigator, Hege Grindem, Associate Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 329-130324
Record Dates: First submitted 2024-05-09; First posted 2024-07-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sports Injury
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The biostatistician performing the main analysis will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- #Utviklingsklar (Experimental): The intervention consists of 1) an e-learning course, 2) a workshop to create plans and practices for injury-prevention, 3) a mid-season meeting
  Interventions: Behavioral: #Utviklingsklar
- Control (No Intervention): Practice as usual, which may include other injury-preventive coaching practices

INTERVENTIONS:
Behavioral: #Utviklingsklar — The intervention consists of 1) an e-learning course, 2) a workshop to create plans and practices for injury-prevention, 3) a mid-season meeting
  Arms: #Utviklingsklar

SUMMARY:
The majority of injuries among Norwegian youth occur in sports. The purpose of the project is to conduct an effect and process evaluation of the intervention #Utviklingsklar, an injury-preventive club-based intervention in youth handball and football. Central to the evaluation is whether the intervention influences the occurrence of new and recurring injuries through changed coaching practices (injury prevention warm-up, strength training, and management of players with pain and injuries). Over one season, participants from 30 clubs in youth handball and football respectively will participate in two cluster-randomized studies. Coaches and club leaders implement #Utviklingsklar and create plans and practices for injury prevention. The control clubs train as usual. Players report injuries. An additional handball and football club are followed up with observation and interviews in a qualitative part of the process evaluation. The project provides knowledge about how injuries and health in the ¾ of Norwegian youth who participate in organized sports are affected by interventions aimed at club and coaching practices.

ELIGIBILITY:
Inclusion criteria:

-Clubs are eligible for participation if they are able to participate with one club leader, 2-6 teams, and a minimum of one coach from each of the participating teams

Exclusion criteria:

* Players under the age of 12
* Coaches under the age of 16

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2954 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-11-09 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Oslo Sports Trauma Research Center Questionnaire on Health Problems (OSTRC-H2) | Average of biweekly reports over 1 sports season (estimated to 32 weeks)
  Weekly injury severity score (0 best - 100 worst)

SECONDARY OUTCOMES:
Sudden and gradual onset injuries | 1 sports season (estimated to 32 weeks)
  Weekly injury severity score during the match season for sudden and gradual onset injuries
Injury location | 1 sports season (estimated to 32 weeks)
  Weekly injury severity score during the match season for lower leg, ankle/foot, knee, shoulder (handball), thigh (football), hip/groin (football), lumbosacral (football) and head (football) injuries
Injury location for sudden onset injuries | 1 sports season (estimated to 32 weeks)
  weekly injury severity score during the match season for sudden onset lower leg, ankle/foot, knee, shoulder (handball), thigh (football), hip/groin (football), and lumbosacral (football) injuries
Injury location gradual onset injuries | 1 sports season (estimated to 32 weeks)
  Weekly injury severity score during the match season for gradual-onset lower leg, ankle/foot, knee, shoulder (handball), thigh (football), hip/groin (football), and lumbosacral (football) injuries
Injury burden | 1 sports season (estimated to 32 weeks)
  Defined as the sum of injury severity score divided by the sum of exposure (per 1000 hours), where the sums are over team and over match season. The unit of analysis for burden is thus team and not player.
Sports Injury Preventive Behavior Questionnaire (construct scores 0 worst - 1 best) | Baseline, midseason and post season (about 32 weeks)
  The aggregated construct scores for the determinants 1) risk perception, 2) intention, 3) outcome expectancies, 4) action self-efficacy, 5) maintenance self-efficacy, 6) coping self-efficacy, 7) recovery self-efficacy, 8) action plans 9) coping plans and 10) club social support
Injury-preventive coaching practices | Baseline and post season (about 32 weeks)
  The injury-preventive coaching practice outcomes consist of:
  1. The change in the extent to which teams complete warm-up as described in the intervention from baseline to end-of season.
  2. The change in the extent to which teams complete strength training as described in the intervention from baseline to end-of season.
  3. The change in the extent to which players with pain or injuries receive guidance on medical care from baseline to end-of season.
  4. The change in the extent to which training and match participation is facilitated for players with pain or injuries from baseline to end-of season.

OTHER OUTCOMES:
Fidelity - workshop completion checklist | At workshop (about 1-2 weeks before sports season)
Fidelity - Midseason meeting checklist | Midseason (about 16 weeks)
Dose - completion of e-learning | Before workshop (about 1-2 weeks before sports season)
Dose - workshop attendance checklist | At workshop (about 1-2 weeks before sports season)
Dose - Midseason meeting checklist | Midseason (about 16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hege Grindem, Principal Investigator — Oslo Sports Trauma Research Center
Locations (6):
- Norway (6):
  - Hordaland Fotballkrets, Bergen
  - Håndballregion Øst, Oslo
  - Oslo Fotballkrets, Oslo
  - Akershus Fotballkrets, Strømmen
  - Håndballregion Nord, Trondheim
  - Trøndelag Fotballkrets, Trondheim

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT06486090/SAP_000.pdf